CLINICAL TRIAL: NCT03969043
Title: Brain Correlates of Visual Processing of Emotional Scenes in ACTion and EMOtional Judgments During Normal VIeillissement
Acronym: ACTEMOVI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Grenoble (Other)
Collaborators: Laboratoire de Psychologie et NeuroCognition (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 38RC18.215; 2018-A02572-53 (Other: ID RCB)
Record Dates: First submitted 2018-12-12; First posted 2019-05-31 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Aging

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Young volunteers (Experimental): Volunteers between 18 ans 45 years old
  Interventions: task scans (n=4), anatomical MRI, Resting state functional scan, Diffusion Tension Imaging, Perfusion imaging.
  Interventions: Other: MRI
- Older Volunteers (Experimental): Volunteers between 60 ans 85 years old
  Interventions: task scans (n=4), anatomical MRI, Resting state functional scan, Diffusion Tension Imaging, Perfusion imaging.
  Interventions: Other: MRI

INTERVENTIONS:
Other: MRI — The MRI examination will consist of a series of acquisition scans:
  * Scanning Scan: for positioning the functional volume of interest.
  * Task Scans: for exploring cerebral activation in emotional and action appraisal tasks during viewing high and low arousal stimuli and a localizer task ".
  * Anatomical MRI: for analyzing the functional images, and measuring volumes of gray and white substances.
  * Resting state functional scan: for exploring cerebral activation during a rest activity.
  * Diffusion Tension Imaging: for measuring structural connectivity.
  * Perfusion imaging: scan for ensuring good perfusion conditions
  All functional acquisitions will be performed in multi-slices in echoplanar mode using gradient echo sequences allowing the exploitation of the BOLD contrast.

SUMMARY:
It is accepted that emotional events engage more attention and are detected and identified faster than neutral events. The same is true of negative events with regard to positive events. At the cerebral level, this facilitation results in greater activation of brain regions involved in visual and emotional processing. In normal aging, the preference for the negative stimuli (named negativity bias) tends to disappear and, sometimes, to shifts towards a preference for positive stimuli compared to both the negative and neutral stimuli (positivity bias). Most studies have assessed the age effect on emotional processing using tasks which require the identification of a personal emotional experience or the emotions of others.

Although many studies suggest a strong link between emotion and action, relatively little is known about the age effect on emotional processing when the task requires the identification of a tendency to action (i.e. preparation of the individual to react and direction of action - example: fear prepares to avoid danger).

ACTEMOVI project aims to identify the brain bases and neural networks involved in the processing of emotional visual information in normal aging when performing emotional appraisal and action-oriented tasks, through a functional MRI study.

DETAILED DESCRIPTION:
It is accepted that emotional events engage more attention and are detected and identified faster than neutral. The same is true for negative events compared to positive events. On the cerebral level, this facilitation results in greater activation of brain regions involved in visual and emotional processing. In normal aging, the preference for the negative stimuli (named negativity bias) tends to disappear and, sometimes, to shifts towards a preference for positive stimuli compared to both the negative and neutral stimuli (positivity bias), which could be mainly related to a decrease with age in processing of negative stimuli and in attention to this type of information. Only a few studies rather suggest an improvement in processing of positive stimuli with age. On the cerebral level, various fMRI studies mainly highlight an age effect on processing of negative stimuli in several brain regions involved in emotional processing such as amygdalae and prefrontal cortex (respectively a lower and higher activity in older adults compared to young adults). This age effect also induces a higher level of well-being and less frequent negative emotional feelings in the elderly than in younger people. Most studies have assessed the age effect on emotional processing using tasks which require the identification of a personal emotional experience or the emotions of others. Although many studies suggest a strong link between emotion and action, relatively little is known about the age effect on emotional processing when the task requires the identification of a tendency-to-action (i.e. preparation of the individual to react and direction of action - example: fear prepares to avoid danger). Team's works on this research question show the negativity bias with age is preserved in a tendency-to-action appraisal task while it disappears with age in an emotional appraisal task, suggesting a dissociation between emotion and tendency to action. In addition, a pilot fMRI study by our team in young people show the tendency-to-action appraisal task compared to emotional appraisal task induces higher activation in brain regions involved in visual and emotional processing. To our knowledge, no study has yet investigated the evolution with aging of neural circuitry involved in emotional processing during a tendency-to-action appraisal task compared to an emotional apparaisal task. Studying this evolution could allow to better understand the observed dissociation with increasing age between emotional and tendency-to-action tasks and more generally to better understand the evolution of the interactions between emotional and action processes with aging.

ACTEMOVI project aims to identify the brain bases and neural networks involved in the processing of emotional visual information in normal aging when performing emotional appraisal and action-oriented tasks, through a functional MRI study and using an original mathematical modeling of functional connectivity based on the Graph theroy developed in the team. Findings will be used to develop a first neural network mapping model involved in visual perception of emotional scenes during emotional and tendency-to-action appraisals during normal aging.

The experiment will be conducted in two age groups (20-35 and 60-85 years old) of 50 healthy participants each (number based on currently requirements in terms of size of effects for the envisaged connectivity analyzes), and carried out using a whole-body 3-T Philips scanner (Philips Medical Systems, Best, NL).

Participants will perform two appraisal tasks during viewing a succession of emotional scenes, one emotional based on the appraisal of personal emotional experience (pleasant, unpleasant or neutral), and the other based on the appraisal of the tendency-to-action (approach, avoidance or no action). Two characteristics of stimuli will be manipulated in the study : valence and arousal.The age effect is modulated by these two characteristics.

For each task, stimuli will be organized into two blocks: "High" block containing pleasant and unpleasant stimuli of high activation and neutral stimuli, and "Low" block including unpleasant and pleasant stimuli of low activation and neutral stimuli. The tendency-to-action induced by stimuli will be congruent with the valence of stimuli (i.e. pleasant/approach, unpleasant/avoidance and neutral/no action). The emotional stimuli in each block will be displayed according to a block fMRI paradigm.

In total, each participant will successively perform four experimental blocks. Two blocks will involve an emotional task (for the high and low blocks) and the other two will involve a tendency-to-action task (for the high and low blocks).The order of tasks and images within a task will be counterbalanced between the participants

For fMRI analyses, the protocol will aso include an anatomical MRI, a Diffusion Tension Imaging (DTI) and a resting-state measure in order to take into account the anatomical and functional differences between age groups. fMRI data (MRI signal of the BOLD type - Blood Oxygen Level Dependent) will be analyzed using standard neuroimaging analysis software (e.g. SPM, FSL). Analysis will perform on whole-body and in regions of interest (ROIs, e.g. amygdala). Regions of interest (ROIs) associated with emotional processing will be functionally identified and delimited for each participant using a separate functional localizer experiment adapted from Vuilleumier et al. (2003). These regions will also be used for Resting-State network analysis.

ELIGIBILITY:
Inclusion Criteria:

* Participant aged between 18 and 45 and between 60 and 85 years old
* Visual acuity normal or corrected to normal
* Affiliation to a social security scheme (copy of the vital card in support)
* Signed informed consent
* Medical examination before taking part in the MRI examination
* Mini-Mental-State Examination Score (MMSE)> 23/30
* Scale score of Beck depression ≤ 4

Exclusion Criteria:

* Participant in other research protocols in progress with exclusion period
* Unprotected Majors unable to express their consent
* Protected Major (Persons mentioned in Articles L1121-5,6 and 8 of the Public Health Code)
* Significant hearing or motor impairment
* Neuropsychiatric or neurological pathology past or present (except benign epilepsy)
* Taking narcotics and / or drugs for neurocognitive purposes
* Existence of a severe condition in general (cardiac, respiratory, hematological, renal, hepatic, cancerous)

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2019-05-10 (Actual); Primary Completion 2021-12-03 (Actual); Study Completion 2021-12-03 (Actual)

PRIMARY OUTCOMES:
Brain activations and connectivities involved in the processing of emotional visual information during normal aging when performing emotional assessment and action-to-action tasks. | 2 hours
  Variables measured from functional MRI data:
  * Statistical maps of brain regions activated in the whole brain for different contrasts of interest for each group of participants (young and old)
  * Statistical activation maps on regions of interest such as amygdala for the different contrasts of interest for each group of participants
  * Functional connectivity between brain regions activated in the whole brain on the basis of correlations and on the basis of graph theory, for different contrasts of interest for each group of participants. Functional connectivity analyzes will be coupled with an analysis of structural connectivity based on Voxel morphometric measurements to voxel of anatomical MRI and Diffusion Tension Imaging data to take account of anatomical differences between age groups. The correlation links between functional and structural connectivities will also be evaluated.

CONTACTS AND LOCATIONS:
Overall Officials: Monica BACIU, Principal Investigator — Grenoble Alpes University Hospital; Aurélie Campagne, Study Director — University Grenoble Alps
Locations (1):
- CHU Grenoble-Alpes, Grenoble, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Poncet E, Nicolas G, Guyader N, Moro E, Campagne A. Spatio-temporal attention toward emotional scenes across adulthood. Emotion. 2023 Sep;23(6):1726-1739. doi: 10.1037/emo0000891. Epub 2022 Nov 28. PMID 36441998